CLINICAL TRIAL: NCT03781180
Title: Randomised, Validity and Reliability Study of the Motor Accuracy Test in Turkey, One of the Sensory Integration and Praxis Tests
Brief Title: Validity and Reliability Study of the Motor Accuracy Test
Acronym: VRMAT
Status: Completed | Type: Observational
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Sponsor
Other Study IDs: 0000-0003-1364-9776
Record Dates: First submitted 2018-01-12; First posted 2018-12-19 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Test-Retest Reliability
Keywords: SIPT; Motor Accuracy; Validity; Reliability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Motor Accuracy-Revised Test's validity and reliability in Turkey was studied in this paper.

DETAILED DESCRIPTION:
The study sample group consists of 100 children who are studying in a primary school registered to Hatay Provincial Directorate of National Education. The children's ages range between 6 years and 8 years 11 months.

ELIGIBILITY:
Inclusion Criteria:

* not having any physical, psychological or mental disabilities,
* to be aged between 6 years and 8 years and 11 months,
* to have the consent of both the child and the parents.

Exclusion Criteria:

* identified as having any kind of physical, visual or hearing disabilities,
* having mental retardation, or possessing a learning disability.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study sample group consists of 100 children who are studying in a primary school registered to Hatay Provincial Directorate of National Education. The children's ages range between 6 years and 8 years 11 months.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Motor Accuracy-Revised Test | 2-weeks
  The Motor Accuracy-Revised Test was implemented on each of the studied children through test-retest.

CONTACTS AND LOCATIONS:
Overall Officials: Fehime S Akbay, MS, Study Director — Academic Member; Ferda Dokuztuğ Üçsular, Professor, Study Chair — Academic Member; Tomris Duymaz, Assist prof, Principal Investigator — Academic Member